CLINICAL TRIAL: NCT00085579
Title: A Phase II Study of Maintenance Biotherapy With Interleukin-2 and Granulocyte-Macrophage Colony Stimulating Factor in Patients With Metastatic Melanoma With a Partial Response or Stable Disease After Systemic Therapy
Brief Title: Interleukin-2 and Sargramostim After Chemotherapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 04-027; MSKCC-04027
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; sargramostim; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: sargramostim
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Interleukin-2 and sargramostim may stimulate a person's white blood cells to kill melanoma cells.

PURPOSE: This phase II trial is studying how well giving interleukin-2 together with sargramostim works in treating patients with stage III or stage IV melanoma that was previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the frequency of complete response in patients with stage III or IV melanoma who have achieved either a partial response or stable disease after prior systemic chemotherapy and are treated with maintenance biotherapy comprising interleukin-2 and sargramostim (GM-CSF).

Secondary

* Determine the time to progression in patients treated with this regimen.
* Determine the effects of this regimen on lymphocyte subsets in these patients.

OUTLINE: Patients are stratified according to response to prior systemic chemotherapy (stable disease [SD] vs partial response [PR]).

Patients receive sargramostim (GM-CSF) subcutaneously (SC) on days 1-14 and low-dose interleukin-2 (IL-2) SC on days 1-5, 8-12, 15-19, and 22-26. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive pulses of high-dose IL-2* IV continuously over 42 hours on days 1 and 2 of courses 2, 3, 5, 6, 8, 10 and 12.

NOTE: *Low-dose IL-2 and GM-CSF are not administered on days 1 and 2 of high-dose IL-2 administration

Patients who continue to have SD or a PR after 12 courses of therapy may continue to receive treatment with GM-CSF and low-dose IL-2 as described above and high-dose IL-2 on days 1 and 2 of every third course.

PROJECTED ACCRUAL: A total of 20-58 patients (10-29 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Stage III or IV disease
  * No primary ocular melanoma
* Stable disease (SD) or partial response (PR) after prior systemic chemotherapy completed at least 4 weeks ago

  * Patients whose second post-chemotherapy evaluation (performed at least 4 weeks after the first evaluation that demonstrated SD or PR AND within 2 weeks before study entry) of disease demonstrates continued tumor shrinkage are not eligible
  * Patients whose second evaluation shows disease progression are eligible unless one of the following is true:

    * Lactic dehydrogenase (LDH) ≥ 2 times upper limit of normal (ULN)
    * LDH > ULN AND is higher than the patient's highest value before systemic chemotherapy
    * Patient has developed a new tumor measuring > 1 cm in diameter
    * Sum of the longest diameters of the existing tumor has increased > 20%
* Evaluable or measurable disease
* Not potentially curable by surgery
* No active CNS metastases

  * Solitary brain metastasis allowed if completely resected or completely ablated with radiosurgery more than 1 month before study entry

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* No active bleeding

Hepatic

* See Disease Characteristics
* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 1.2 mg/dL

Cardiovascular

* Patients ≥ 50 years of age OR those with one or more cardiac risk factors must demonstrate one of the following:

  * Normal exercise stress test
  * Normal stress thallium test
  * Normal comparable cardiac ischemia evaluation
* LVEF ≥ 40%

Other

* No active infection requiring treatment
* No concurrent medical or psychiatric condition that would increase the potential toxicity of study treatment
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent antineoplastic biologic response modifier therapy
* No concurrent antineoplastic vaccine therapy

Chemotherapy

* See Disease Characteristics
* No concurrent antineoplastic chemotherapy

Endocrine therapy

* No concurrent steroidal antiemetics
* No concurrent systemic corticosteroids

Radiotherapy

* See Disease Characteristics
* No concurrent antineoplastic radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery
* Surgery within the past 4 weeks allowed provided there is no evidence of disease progression

Other

* More than 4 weeks since prior therapy for melanoma
* No other concurrent antineoplastic experimental therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Jedd D. Wolchok, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States